CLINICAL TRIAL: NCT02388542
Title: Policy and Peer Mentor Intervention Programs on Cardiovascular Disease at Small to Medium Sized Worksites in 3 South Asian Countries - a Pilot Study for a Definitive Large International Cluster Randomized Trial
Brief Title: Effect of Peer-mentor Mediated Interventions on Cardiovascular Risk Factors at Worksites
Acronym: PROGRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. John's Research Institute (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Colombo (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PROGRESS-IND-1022015
Record Dates: First submitted 2015-02-09; First posted 2015-03-17 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2016-10

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular disease; education; peer mentor
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counseling (Experimental): we will have a trained peer mentor educating employees regarding lifestyle modification for control of cardiovascular disease risk factors and following them up for a duration of 3 months
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — Employees above the age of 35 years will be risk stratified into moderate or high risk of developing cardiovascular disease using a simple non-lab based risk scoring system, they will be invited to participate in the pilot intervention study. This is a single arm before-after study.subject education will focus on life style medication and adherence to medication (if applicable).importantly the peer mentor will try to identify barriers to adopting a healthy lifestyle(tobacco, physical acitivity, diet, alcohol and strees) and adherence to cardiovascular disease prevention medication. peer mentors will be trained to interpret blood glucose and lipids, recognize abnormal valves, provide lifestyle counseling and refer to treating physician when appropriate.

SUMMARY:
The investigators propose conducting a pilot study to identify 6 worksites (2 India, 2 Sri Lanka, 2 Bangladesh) explore barriers to optimum cardiovascular disease(CVD) care at these worksites, quantify risk factor level in worksite populations and identify and train peer mentors to deliver an educational intervention to improve life style and enhance medication adherence among those at moderate to high risk of cardiovascular disease (CVD).

DETAILED DESCRIPTION:
Eligibility Criteria -

All employees aged above 35 years at selected workplaces.

Study design - Mixed methods methods Phase 1 - Qualitative study; Phase 2 - Quantitative - Single group, non-randomized before-after comparison study + KAP survey

Sample size - Approximately 334 participants.

The study entails the following steps -

Step 1 - An evaluation for knowledge, attitudes and practices (KAP) related to cardiovascular health/ disease at worksites.

Step 2 - A qualitative study for barriers and facilitators of behaviors associated with optimal cardiovascular health

Step 3 - Baseline assessment of cardiovascular risk using a non-lab based risk assessment score

Step 4 - Piloting a trained peer mentored educational/ intensive follow-up intervention for 3 month with a re-assessment at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* All criteria must be met to be eligible

  1. Employees (Men & Women) above the age of 35 years.
  2. permanent employees with at least 6 months for retirement.
  3. Willing to provide Informed Consent.

Exclusion Criteria:

* Subject ineligible if even one criterion is met

  1. Pregnant or intent to get pregnant in one year.
  2. Inability to attend follow up visits.
  3. Any active malignancy or known malignancy on treatment.
  4. Will relocate during the study period.
  5. Unwilling or unable to comply with study procedures.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge attitudes & practices related to Cardiovascular risk factors. (questionnaire) | 1 Month
  A knowledge, attitudes & practices questionnaire will be administered to participants
Identification of barriers and facilitators for an optimal Cardiovascular Health environment. (In depth interviews and focus groups discussions with random sample of participants) | 3 Months
  qualitative analysis - In depth interviews and focus groups discussions with random sample of participants
Estimate the Cardiovascular risk factor burden (validated non lab based Cardiovascular risk score) | 3 Months
  validated non lab based Cardiovascular risk score will be used (developed from NHANES data and validated against Framingham score

CONTACTS AND LOCATIONS:
Overall Officials: Dr Denis Xavier, M.D,MSc., Principal Investigator — St.John's Medical College
Locations (6):
- Bangladesh (2):
  - Appollo Ispat Complex Ltd, Dhaka
  - Shardharan Bima Coorporation, Dhaka
- India (2):
  - Bharat Heavy Electrical Limited, Bangalore
  - TVS Motor company Limited, Hosūr
- Sri Lanka (2):
  - Department of Census & Statistics, Colombo
  - Sri Lanka Telecom, Colombo